CLINICAL TRIAL: NCT05815914
Title: Dietetic Education Support, and Nutrition to Chronic Complex Patients With the Usage of a Telemedicine Tool
Brief Title: Nutritional Support and Telemedicine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20/92
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Malnutrition
Keywords: Telemedicine; nutritional support; polimorbidity patients
MeSH Terms: conditions — Malnutrition | interventions — Amyloid; Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: app
- Control group (Active Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: app — The app will include a nutritional education programme through the APP throughout the study. At 2, 4, 6 and 8 months data will be collected through a telematics questionnaire
  Arms: Intervention group
Other: control group — Routine nutritional and dietary recommendations will be given.
  Arms: Control group

SUMMARY:
The aim of this clinical trial is to assess the implementation of an APP to track the nutritional status and diet habits of "chronic complex patients"(CCP) in order to improve their nutritional status and evaluate the level of adherence to dietetic counseling.

DETAILED DESCRIPTION:
The aim is to evaluate the usage of an APP and track the nutritional status of "chronic complex patients"(CCP) in order to improve their nutritional status.

This is a study of an experimental design, referring to a controlled randomized trial with CCP in the Moises Broggi hospital.In the first stage, there's been an elaboration of the contents of the APP. For the assessment of the strategy of food education, two groups of patients will be defined(Intervention group (IG) & Control group (CG)). In each group there will be 91 subjects, meaning a total of 182 patients. Inclusion criteria: >18 years old, CCP with either malnutrition, or risk of malnutrition (MNA<23,5), therapeutic profile <3, living at home, with full accessibility and capable to use a smartphone, and usual internet consumers (patients or caregivers), and who need to sign the informative consent. The inclusion of this study, will be made through a random sampling and patients will be assigned to IG or CG. All patients will undergo an initial evaluation, a follow-up visit after the first 6 months, and then a final visit after 12 months. The intervention group will also contain an educational, and nutritional program by means of the APP throughout the entire study, and data will be collected through a telematic questionnaire between visits. The variables to study are nutritional, diet, clinics, social and valorisation tools ICT (IG).

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* polymorbidity
* malnourished patient or patient at risk of malnutrition (MNA≤23.5)
* patient living at home, with access to and able to use a smartphone and regular internet users (patients or caregivers)
* patient who agrees to participate in the study by signing the informed consent form

Exclusion Criteria:

* established artificial nutrition
* advanced dementia
* admission to a nursing home/social care for a period of >1 month
* patients not responding to the telematic visits on more than 2 occasions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in nutritional status | Baseline and 12 months
  Assessment of changes in nutritional status through the Mini Nutrition Assessment (MNA) at baseline and at 12 months

SECONDARY OUTCOMES:
Adherence to the Mediterranean diet | 12 months
  Assessment of adherence to the Mediterranean diet will be carried out with by Predimed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Sant Joan Despí, CSI, Sant Joan Despí, Barcelona, Spain